CLINICAL TRIAL: NCT04866082
Title: Administration of Systemic Corticosteroids Among Critically Ill Patients With COVID-19: Electronic Survey Within European Society of Intensive Care (ESICM) and European Society of Anaesthesiology and Intensive Care Members (ASAP-ESICM/ESAIC Study)
Brief Title: Corticosteroids in Severe COVID-19 (ASAP-ESICM/ESAIC Study)
Acronym: ASAPESICMESAIC
Status: Completed | Type: Observational
Sponsor: Brno University Hospital (Other)
Collaborators: European Society of Intensive Care Medicine (Other); European Society of Anaesthesiology and Intensive Care (Other)
Responsible Party: Principal Investigator, Jan Malaska, assoc.prof.MD,Ph.D, Brno University Hospital
Other Study IDs: ASAP-ESICM/ESAIC
Record Dates: First submitted 2021-04-26; First posted 2021-04-29 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Severe COVID-19
Keywords: COVID-19; ARDS; corticosteroids; critical care
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ESICM and ESAIC members: questionnaire - Members of European Society of Intensive Care and European Society of Anaesthesiology and Intensive Care will obtain an electronic survey regarding their routine clinical practice of systemic corticosteroids administration among patients with COVID-19 ARDS
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — Members of European Society of Intensive Care and European Society of ANaesthesiology and Intensive care will obtain an electronic survey regarding their routine clinical practice of systemic corticosteroids administration among patients with COVID-19 ARDS
  Other Names: electronic survey

SUMMARY:
Brief Summary: Administration of systemic corticosteroids for patients with severe forms of severe acute respiratory syndrome in coronavirus-2 (SARS-CoV-2) infection are recommended by several guidelines. In the very beginning of SARS-CoV-2 pandemic the early recommendation by professional organization was against routine use of corticosteroids for patients with coronavirus disease 2019 (COVID-19) ARDS, despite previous data and clinical practice for patients with refractory or severe form of acute respiratory distress syndrome (ARDS). But recently after publication of RECOVERY trial (Randomized Evaluation of Covid-19 Therapy, July 2020) and ensued metaanalysis of World Health Organization (WHO) working group, routine administration of systemic corticosteroids was revisited. However, there is an ongoing debate regarding evidence supporting the dose, type of administration (bolus vs. continuous infusion), timing and type of corticosteroids. Ongoing randomized controlled trials (RCTs) are challenging the recommendation of 6 mg of dexamethasone for all patients with severe form of COVID-19. Due to the dynamics of COVID-19 surges and rapid issuing of official recommendations, daily clinical practice of systemic corticosteroids administration can vary. An electronic evaluation form containing 20 questions will be sent to European Society of Intensive Care (ESICM) and European Society of Anaesthesiology and Intensive Care (ESAIC) members. Participants will be asked to describe their routine clinical practice regarding administration of systemic corticosteroids among patients with COVID-19 ARDS.

DETAILED DESCRIPTION:
Brief Summary: Administration of systemic corticosteroids for patients with severe forms of SARS-CoV-2 infection are recommended by several guidelines. In the very beginning of SARS-CoV-2 pandemic the early recommendation by professional organization was against routine use of corticosteroids for patients with coronavirus disease 2019 (COVID-19) ARDS, despite previous data and clinical practice for patients with refractory or severe form of ARDS. But recently after publication of RECOVERY trial (Randomized Evaluation of Covid-19 Therapy, July 2020) and ensued metaanalysis of WHO working group, routine administration of systemic corticosteroids was revisited. However, there is an ongoing debate regarding evidence supporting the dose, type of administration (bolus vs. continuous infusion), timing and type of corticosteroids. Ongoing RCTs (Randomized Clinical Trials) are challenging the recommendation of 6 mg of dexamethasone for all patients with severe form of COVID-19. Due to the dynamics of COVID-19 surges and rapid issuing of official recommendations, daily clinical practice of systemic corticosteroids administration can vary. An electronic evaluation form containing 20 questions will be sent to European Society of Intensive Care (ESICM) European Society of Anaesthesiology and Intensive Care (ESAIC) members. Participants will be asked to describe their routine clinical practice regarding administration of systemic corticosteroids among patients with COVID-19 ARDS.

ELIGIBILITY:
Inclusion Criteria:

* Members of European Society of Intensive Care (ESICM)
* Members of European Society of Anaesthesiology and Intensive Care (ESAIC)

Exclusion Criteria:

* not members of European Society of Intensive Care (ESICM)
* not members of European Society of Anaesthesiology and Intensive Care (ESAIC)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Members of European Society of Intensive Care Members of European Society of Anaesthesiology and Intensive Care (ESAIC)
Sampling Method: Non-Probability Sample
Enrollment: 466 (Actual)
Dates: Start 2021-05-30 (Actual); Primary Completion 2022-06-14 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Administration of systemic corticosteroids among patients with COVID-19 ARDS practice in European countries - questionnaire (electronic survey) | 2 months
  Electronic survey will be send to the European Society of intensive care (ESICM) members via email

CONTACTS AND LOCATIONS:
Overall Officials: Jan Malaska, assoc. prof. MD., Ph.D., Study Director — University Hospital Brno; Petr Stourac, prof.MD.Ph.D., Study Chair — Faculty of medicince Masaryk University and University Hospital Brno
Locations (1):
- Brno University Hospital, Brno, South Moravian, Czechia

IPD SHARING:
Plan to Share IPD: Undecided